## A Phase II Biomarker Trial of Avadomide (CC-122) in combination with Nivolumab in Advanced Melanoma

# NCT03834623 ICF Version 3 Dated 12/06/2019

## CONSENT TO TAKE PART IN A CLINICAL RESEARCH STUDY AND AUTHORIZATION TO DISCLOSE HEALTH INFORMATION

Study Title: A Phase II Biomarker Trial of Avadomide (CC-122) in

combination with Nivolumab in Advanced Melanoma

Protocol Number: MCC 19706

Sponsor: Moffitt Cancer Center

Principal Investigator:

(Study Doctor)

Nikhil Khushalani, MD

Telephone: (813) 745-3437 (24 hour number) (800) 456-3434

Address: Moffitt Cancer Center McKinley

10920 N. McKinley Tampa, FL 33612

Moffitt Cancer Center 12902 Magnolia Drive Tampa, FL 33612

This consent and authorization form explains why this research study is being done and what your role will be if you choose to take part. You may choose not to take part in this study.

The purpose of this study is to find out if the combination of Avadomide (CC-122, an investigational agent) and Nivolumab will result in improved anti-cancer activity and prevent T-cell exhaustion (T-cells are responsible for maintaining your body immune response) in your advanced melanoma condition. This is a type of skin cancer, but this has now spread to other organs, and cannot be removed by surgery.

The researchers will look for early signals that the study treatment is working (for example, tumor shrinkage, survival rate) and want to learn about the tolerability and toxicity of this combination.

Another purpose of the study is to learn more about how the compounds work in combination, to get an early picture of what they do to biomarkers (for example, proteins) in the blood and tumor, and if these biomarkers in blood and tumor change over the course of the study. Biomarkers are substances in the body that increase or decrease in expected ways following study treatment. Studying these biomarkers while you are receiving study drugs may show



whether or not the study drugs are affecting your tumor. The relationship between the amount of study drug in your body and the effect of the biomarkers on your disease when the study drugs are given as pairs will also be studied.

Your total participation in this study from the time you sign and date the informed consent form through your last visit may be up to about 36 months, depending on how your cancer responds to the study treatment and depending on your test results.

Before you can start the study, the study doctor or study staff will talk to you about the study. If you agree to participate, you have to sign and date this form before the study doctor or study staff can begin the first part of the study called a screening period (for a period of up to 28 days) to see if you qualify to be in the main part of the study. Your study doctor will determine your eligibility to participate in the study. If you qualify to continue in the study you will undergo a study treatment visit. This will involve administration of the investigational drug along with other study procedures which are later described in detail in this document. Post-study treatment visit, you will have an end of study treatment/follow-up visit which involves evaluating your health condition by routine clinic examination and procedures, later described in detail. Your regular medical care might include some of the study tests and procedures. The study doctor or a member of the study staff can answer any questions you may have about which tests and procedures are not part of your regular medical care

We anticipate enrolling between 44 to 66 participants in this study at Moffitt Cancer Center. Your participation is voluntary, and you may stop your participation at any time. There will be no penalties or loss of benefits or opportunities if you do not participate or decide to stop once you start.

Alternatives to participating in the study include – getting treatment or care for your cancer without being in a study (typically called standard of care treatment), taking part in another study of an investigational drug, and getting no treatment.

If you decide that you don't want any more active treatment, one of your options is called "comfort care", also called palliative care. This type of care aims to help reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible. If you think you might prefer comfort care, please discuss this with your family, friends and your study doctor. Talk to your study doctor about your choices and the risks and benefits before you decide if you will take part in this study.

We do not know if you will receive any benefit from your participation. You will not be compensated for your participation.

The most common and most serious risks that may be related to Avadomide includes fatigue, weakness, low blood counts, decreased appetite, nausea, vomiting, diarrhea, constipation, rash, fever, infection. The most common risks due to Nivolumab include diarrhea, fatigue, itching and rash. The other risks and side-effects due to use of investigational drug and risks associated with other study procedures are described later in this consent form.

Any new important information that is discovered during the study and which may influence your willingness to continue participation in the study will be provided to you.

Even if we publish the findings from this study, we will keep your study information private and confidential. Anyone with the authority to look at your records must keep them confidential.

If you are interested in learning more about this study, please continue reading the information below:

#### WHAT IS THIS STUDY ABOUT?

We are asking you to take part in this research study because you have been diagnosed with 'unresectable or metastatic melanoma' (one of the types of skin cancer). This disease condition means that your skin cancer has spread locally or to other organs and cannot be removed or is unresponsive to surgical treatment.

Your study doctor considered you as a potential participant because you are treatment naïve for the present stage of your cancer (meaning you would be receiving study treatment for the first time) or you were treated with the study drug in the past and then your symptoms returned during therapy or after discontinuation of study drug.

In this study, you will be treated with an investigational drug called Avadomide. The use of Avadomide is experimental. An "investigational drug" is a drug that is being tested and is not approved for sale in the United States by the U.S. Food and Drug Administration (FDA).

Avadomide (CC-122) is manufactured by Celgene Corporation. It is a drug that has not been approved in any country for the treatment of any medical condition and is investigational (being tested) in this study. It is a "pleiotropic pathway modulator" that may affect cancer in many ways. Pleiotropy refers to a case where one target may influence several other characteristics or may have multiple effects in numerous tissues such as tumor, blood vessels and cells of the immune system. Avadomide comes in capsules that are taken by mouth and swallowed with water. It is being studied as a possible treatment for advanced solid (organ) tumors, non-Hodgkin's lymphoma, chronic lymphocytic leukemia, and multiple myeloma (a type of blood cancer).

Nivolumab (Anti PD-1) (OPDIVO®) is an antibody (a type of human protein) already approved by the FDA for the treatment of melanoma and several other cancers including metastatic kidney carcinoma, urothelial carcinoma, non-small cell and small cell lung cancer, squamous cell carcinoma of the head and neck, hepatocellular (liver) carcinoma, Hodgkin's lymphoma, selected colon cancers, and cancers with high microsatellite instability (MSI-H). Nivolumab (Anti-PD-1 inhibitor) is effective in reducing the tumor induced immune suppression and can be given by itself or in combination with another drug called ipilimumab for the treatment of advanced melanoma based on current approval by the FDA in the United States. In melanoma, it is also approved after surgery to reduce the risk of recurrence in patients with stage III (lymph node involvement) or stage IV disease who have had all their cancer removed by surgery.

#### WHAT WILL HAPPEN DURING THIS STUDY?

Your study participation is divided into a Screening period, a Study Treatment period (each cycle for 28 days with Day 1 and Day 15 visits at the study doctor's office for Nivolumab administration and other study procedures), and End of Study Treatment period.

#### **Screening Period**

Before you begin any part of this study, you must sign and date this consent form. You must be honest with your study doctor about your health history and medication use or it may not be safe for you to be in this study. If you decide to take part in the study, your study doctor must be sure that you are well enough to undergo the study treatment. This screening examination will involve:

- Physical Exam including your height and weight
- Medical History/Oncology History including questions regarding tobacco and alcoholuse
- Vital Signs (blood pressure, heart rate, and temperature)
- Pregnancy Test blood (only for women who are able to get pregnant)
- Hormonal blood tests to assess your thyroid and adrenal gland function
- Testosterone Test blood (only for men)
- Blood tests to monitor your general health
- Performance status evaluation (what type of daily activities you can do)
- Blood for biomarker testing and other study procedures.
- If you are eligible to participate in this study, you will undergo one or more of the study procedures described in this form at each study visit

#### **Study Treatment Period**

Each study treatment cycle is 28 days long. When you complete the study treatment or stop the study treatment for any reason, you will have an end of study treatment visit before entering the follow-up period.

When you return for your Cycle 1 Day 1 visit, you will have the following procedures:

- Physical Exam
- Weight
- Vital Signs (blood pressure, heart rate, and temperature)
- Pregnancy test: blood (only for females who are able to get pregnant
- Demographic and medical history
- Blood tests to monitor your health
- Performance status evaluation
- Blood for biomarker testing and other study procedures.

On Day 1 of each study treatment cycle, during your study doctor visit, you will first receive Avadomide to take by mouth. You will receive a fixed dose of Nivolumab by a needle inserted into your vein (IV). On Day 2 through Day 5 of the study treatment cycle, you will take Avadomide at home. Try to take it in the morning and at about the same time that you took them on Day 1. On Day 6 through Day 7 of the study treatment cycle, no study drug will be taken. On Day 8 through Day 12 of the study treatment cycle, you will only take Avadomide capsule(s) at home. On Day 13 through Day 14 of the study treatment cycle, no study drug will be taken. On Day 15, you will return to your study doctors' office for the Cycle 1 Day 15 visit.

On the Cycle 1 Day 15 Visit, the following set of procedures will be performed:

- Physical Exam
- Weight
- Vital Signs (blood pressure, heart rate, and temperature)
- Pregnancy test: blood (only for women who are able to get pregnant)
- Demographic and medical history
- Blood tests to monitor your health
- Performance status evaluation
- Receive another 240mg IV infusion of Nivolumab
- Blood for biomarker testing and other study procedures

On Day 15 through Day 19 of the study treatment cycle, you will only take Avadomide capsule(s) at home. On Day 20 through Day 21 of the study treatment cycle, no study drug will be taken. On Day 22 through Day 26 of the study treatment cycle, you will only take Avadomide capsule(s) at home. On Day 27 through Day 28 of the study treatment cycle, no study drug will be taken. Your study doctor or his/her study staff will give you clear instructions for taking study drugs. This way you will complete your Cycle 1 (28 days).

Between Days 22 and 29, a tumor biopsy will be repeated from the same site where the prestudy treatment biopsy was taken.

After completing 28 days in your Cycle 1, you will return to study doctor for your Cycle 2 Day 1 and other subsequent study treatment visit which will follow the same 28-day cycle. You can refer the 'Schedule of events' calendar included in this document and discuss with your study doctors and study staff for any questions about study related procedures.

#### **End of Study Treatment Period**

This visit starts when your study treatment is completed, changed or discontinued for any reason. The visit will be within 30 days after you complete or stop the study treatment.

- Medical History
- Weight
- Physical Examination
- Tumor Measurement
- Vital Signs (blood pressure, heart rate, and temperature)
- Demographic and medical history
- Blood tests to monitor your health
- Performance status evaluation
- Blood for biomarker testing and other study procedures
- Optional tumor biopsy

If your study discontinuation is due to some study related toxicity or adverse event (bad side effect), you will be followed up until the adverse event is resolved.

If you discontinue the study treatment for a reason other than disease progression or disease-related toxicity, your study doctor will assess your condition every 12 weeks by radiology imaging techniques (computed tomography [CT] scan, magnetic resonance imaging [MRI] scan, positron emission tomography [PET] scan) to monitor your condition for up to 24 months.

If your melanoma responds well to the study treatment, your study doctor will use these follow-up visits to make sure it continues to do well. If the study treatment does not work as expected or stops working, your study doctor will use future follow-up visits to ask some questions about how you are doing and what other treatments you are receiving for melanoma. These questions can be asked over the telephone and you will not need to come to the study doctor's office for a visit.

The maximum time you will be in the study depends on many factors like how your melanoma responds to the study treatment, and how long the study has been open when you join.

The study doctor or study staff will do the things listed below when you come in for study visits. If you would like more information about which tests and procedures will be done at each study visit, ask the study doctor or study staff.

**Medical History:** Will be checked on screening visit, Cycle 1 Day 1, Cycle Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3, other subsequent visits and the end of study treatment visit. The study doctor will ask you about past/present diseases and surgeries. The questions may also include any allergies, birth control procedures and medicines. Any other studies you were in may also be asked. Other questions may include any medical conditions or side effects which may occur during the study.

**Vital Signs, Height and Weight:** Will be checked on screening visit, Cycle 1 Day 1, Cycle Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3, other subsequent visits and the end of study treatment visit. Check your blood pressure by putting a band around your arm (this will squeeze your arm for about a minute), check your pulse, listen to you breathe in and out, and take your temperature. Body weight is also recorded to see how much you weigh.

**Demographic Data**: At Screening, demographic information like your year of birth, gender, and ethnic origin will be collected if permitted by local regulations.

**Physical examination**: Including symptoms of your disease will be performed at Screening, prior to receiving study treatment on Day 1 and Day 15 of each study treatment cycle, at the end of study treatment visit and at each follow-up assessment.

**Concomitant Medication:** You will be asked about the medications you take currently and any medication prohibited taking while on the study. This will be asked at Screening, and on Day 1 of each study treatment cycle.

**ECOG** (Eastern Cooperative Oncology Group) Performance Status: This is a scale used by doctors to describe how well a cancer patient is able to function. It assesses the patient's ability to do daily activities like bathing and getting around. Your ECOG performance status will be assessed at Screening, on Day 1 of each study treatment cycle, at the end of study treatment and at the 28-day follow-up visit.

**Study Diary:** You will be given a study diary to assess compliance with Avadomide therapy. You will be asked to mark on a paper 'diary card' each time you take your doses of Avadomide. You will bring the diary card with you to your next study doctor's visit. You must bring your bottle of study drug (even if empty) with your diary to all your scheduled study doctor visits.

**Tumor Biopsy/Core Needle Biopsy:** Tumor biopsies will be done before study treatment during the screening period, between Day 22 and Day 29 of Cycle 1, and in some cases at the end of study treatment visit (if your cancer is no longer responding to the study treatment; your study doctor will discuss this with you to see if you are willing to participate in this). These biopsies will be either core needle biopsies (or punch biopsies if skin lesions) depending on which type your study doctor thinks will be possible on your tumor. Additional optional biopsies may be done with your permission.

**Echocardiogram (ECHO) or multiple gated acquisition scan (MUGA):** This shows how well your heart is beating and pumping blood and if there are abnormalities present. This will be performed at Screening visit and Day 1 of Cycle 3. This test is a study requirement and usually not part of your routine cancer care.

**Pregnancy Testing:** You will have either a blood pregnancy test (1 teaspoon or 5 milliliters) during the screening period prior to beginning the study treatment and on Day 1 of each cycle of study treatment. Women who are able to become pregnant must agree to use two effective birth control methods (for example: birth control pills, condoms) at the same time or practice

complete abstinence from sexual contact with a man beginning 28 days before starting study treatment, throughout the entire duration of study treatment including, during any dose interruptions, and for at least 28 days after the end of study treatment with Avadomide. Please see risk section below for additional birth control requirements.

**Testosterone testing:** For male participants only, will be done only at Screening.

**Tumor Measurement:** Your tumor will be measured every 12 weeks unless your disease shows progression and you are taken off study based on standard imaging criteria. The imaging is considered standard of care.

- Computed tomography (CT) scan is a type of X-ray scan. Several X-rays from different angles are sent through the body at one time. A computer processes the results to give a better picture than a standard, single X-ray scan. Also, a special dye is used to help improve the picture quality. The dye that is injected into your body may cause you to get a metallic taste in your mouth and to feel warm. Rarely, it causes nausea and vomiting. The dye can also cause damage to the kidneys, which may lead to kidney failure. This is a concern if you have poor kidney function. Rarely, the dye can cause a life threatening reaction. The results are shown as a flat picture (length and width) displayed on a computer screen. Your neck, chest, stomach area, and pelvic/hip area will be scanned. A small amount of dye is inserted into your vein just before the pictures are taken. CT scans will be performed at Screening and every 12 weeks. This is the preferred method to follow the progress of your cancer.
- Positron emission tomography (PET) scan is a type of X-ray scan that uses a radiotracer called fludeoxyglucose (FDG). The tracer is a sugar that carries a small amount of radiation and helps improve the picture quality. Importantly, the FDG tracer shows how fast a tumor is growing. The results are shown as a 3D picture (length, width, and depth) displayed on a computer screen. Your neck, chest, stomach area, and pelvic/hip area will be scanned. A small amount of tracer is inserted into your vein just before the pictures are taken. PET will be done at Screening and every 12 weeks. This will be done only if you have specific reasons not to undergo a contrast CT scan to follow the progress of your cancer.
- Magnetic resonance imaging (MRI) scan: An MRI machine or scanner uses a strong magnet and radio waves connected to a computer to create pictures of parts of the body. In this study, you will have an MRI of your brain. The MRI unit is a large magnet that looks like a donut. A sliding table is in the opening. You will lie on the table and be comfortably positioned. In many cases, an extra piece of imaging equipment called a coil will be placed over the area of your body that is being imaged. The table will move into the opening. The technologist will be just outside the scanner room, but can see, hear, and speak to you at all times. During the exam, you will need to remain very still. Being in a tight enclosed space may make you feel anxious.

**Blood samples:** To check your blood cell counts, heart, liver, and kidney function and other standard safety tests during study treatment. About 2 to 4 tablespoons or 30 to 60 milliliters of blood will be taken per test day. Blood samples are taken at Screening, on Day 1 and Day 15 of each study treatment cycle and at the end of study treatment.

**Thyroid Stimulating Hormone (TSH) test:** To check the function of your thyroid gland during study treatment. Blood samples are taken at Screening, and on Day 1 of Cycle 2 and Cycle 3 study treatment.

**Troponin and Brain Natriuretic Peptide (BNP) test:** To monitor for possible early signs of damage to your heart. Test will be performed at Screening and on Day 1 of every study treatment cycle.

**Biomarker Sampling:** To check the effect of study treatment, blood will be taken for biomarker testing. The blood samples will be taken for biomarker analysis on the following days: Screening, Day 1 and Day 15 of Cycles 1 and 2, and at selected time points thereafter.

#### **Study Treatments**

If you meet eligibility criteria, you will be assigned to receive Avadomide (CC-122) and Nivolumab during this study.

Nivolumab (240mg IV): This drug is administered by intravenous (IV) infusion, meaning the study drug is a solution given through a vein. A pump will be used to ensure correct amount of study is given over the proper amount of time. The infusions can take about 30 minutes per visit.

| Study Drug | Infusion Time | Frequency | Study Treatment Duration |
|---|---|---|---|
| Nivolumab (240 mg) | 30 minutes | Every 2 weeks (Day<br>1 and Day 15 of each<br>cycle) | Up to 52 weeks<br>(about 26 doses) |

If your cancer is continuing to show improvement at the 52-week mark, you will be given the option of continuing study treatment.

<u>Avadomide (CC-122):</u> Avadomide comes in capsules that should be stored as directed on the label. In this study, this study will be available in 3 different doses. You drug dose will be adjusted if you experience any toxicity at the given dose, and your study doctor will make that determination

| Avadomide | Dose and schedule: 5 days on, 2 days off |
|---|---|
| Starting dose | 2 mg |
| 1 <sup>st</sup> Dose Reduction | 1.5mg |
| 2 <sup>nd</sup> Dose Reduction | 1 mg |

On Day 1 of each 28-day study treatment cycle, you will receive 2mg of Avadomide while you are at the study doctor's office, before receiving Nivolumab. Avadomide is taken for 5 days each week, followed by 2 days without taking Avadomide (5/7 days). Your study doctor or his/her study staff will give you clear instructions for taking Avadomide.

On most days, you will take your dose of Avadomide at home. You will be asked to mark on a paper 'diary card' each time you take your dose of Avadomide. You will bring the diary card with you to your next study doctor's visit. Once at home, you should take Avadomide with plenty of water at about the same time on every dosing day. If you forget to take a dose of Avadomide you can take it up to 12 hours later on the same day. If you are late by more than 12 hours, you should not take Avadomide that day, and take your next dose as planned. If you ever have questions about how to take your study drug, you should call your study doctor.

You must bring your bottle of study drug (even if empty) with you to all your scheduled study doctor visits.

You may continue taking Avadomide until:

- You have completed study treatment,
- Your disease gets worse,
- You have a serious side effect that is not tolerated, or
- You or your study doctor decides to stop study treatment for any reason.

#### **Schedule of Event Calendar**

| | Pre-<br>study/Screening | C1D1 | C1D15 | C2D1 | C2D15 | C3 and<br>beyond | End of<br>Study<br>Treatment |
|---|---|---|---|---|---|---|---|
| Informed consent | x | | | | | | |
| Medical history | X | X | X | X | X | X | X |
| Demographics | x | | | | | | |
| Weight | X | X | X | X | X | X | X |
| ECOG Performance status | X | X | | X | | x | x |
| Concomitant medications | X | x | | x | | X | |
| Vital signs | x | X | X | X | X | X | X |
| Physical examination | x | X | x | X | x | x | x |
| Tumor measurement | x | | | | | x | x |
| Blood samples | x | X | X | X | X | X | X |
| Pregnancy test | X | X | | X | | X | |
| TSH | x | | | X | | X | |
| Testosterone (men only) | X | | | | | | |
| Troponin & BNP | x | | | X | | X | |
| Echo / MUGA | x | | | | | X | |
| Blood for Biomarker<br>Analysis | x | x | x | x | x | x | x |
| Nivolumab (240mg IV) | | X | x | X | | | |
| Avadomide (CC-122) | | X | | X | | x | |
| Tissue Biopsy | x | | | x | | | x |

#### WHO IS PAYING FOR THIS STUDY?

A company called Celgene Corporation, the sponsor of the study, is paying for this research study. Avadomide is manufactured by Celgene and will be provided by them to you at no cost.

#### INSTITUTIONAL CONFLICT OF INTEREST MANAGEMENT PLAN

Moffitt Cancer Center, sponsor of this study has a license agreement with Celgene Corporation, company supplying study drug. Payments have been distributed to the Moffitt Cancer Center and Moffitt Cancer Center inventors of the licensed technology which is not a part of this study. The Moffitt Cancer Center and those inventors are also entitled to receive additional payments related to the licensed technology. This study has been carefully reviewed to help assure that the professional judgement of the Moffitt Cancer Center doctors and staff will not be compromised. The study will be monitored for your safety and to ensure the proper analysis of data. Any questions you might have about this study will be answered by Dr. Nikhil Khushalani, the Principal Investigator (the person in charge of this research study), at the telephone number listed on the first page of this document or the Moffitt Cancer Center Compliance Office at (813) 745-1869. Dr. Khushalani does not have a financial relationship with Celgene.

#### WILL IT COST ANYTHING TO BE IN THIS STUDY?

You and/or your insurance company will be financially responsible for hospital inpatient, outpatient and follow-up visits that would normally or routinely occur in the management of your disease. Inpatient and outpatient visits could include charges for treatments, medications, physician visits, laboratory tests and procedures. You and /or your insurance company will be responsible for paying for the charges which are considered routine, since you would have received these services even if you were not participating in this study. You will be responsible for any costs not covered by your insurance company, including deductibles, co-payments and all out-of-pocket expenses. Before you agree to be in this study, you should contact your health insurer to see if your plan will cover the costs required as part of your participation.

You and/or your insurance company will not be responsible for paying for study related items and services that are specifically required for this research study and are not considered part of the routine management of your disease, if these procedures are performed at Moffitt Cancer Center.

During your participation in this study, the study sponsor will be responsible for providing the study drug, CC-122, at no additional charge to you.

You and/or your insurance company will be responsible for the drug nivolumab that is commercially available. You and/or your insurance company will be responsible for the charges related to the administration of the commercially available drugs.

If you would like more information on the costs of being on this study or have other insurance related questions then please let your clinical trial coordinator know or contact our Business Office at 813-745-8422.

#### WILL BEING IN THIS STUDY HELP ME?

If you agree to take part in this study, there may or may not be direct medical benefit to you. Your condition may stay the same or it may get worse during the study. The information collected during this study will help researchers learn more about the study drug combination and may benefit you and other people with melanoma in the future. However, there is no guarantee that this will happen.

#### ARE THERE RISKS TO ME IF I AM IN THIS STUDY?

Right now, we do not know for sure if combination of Avadomide and Nivolumab will help. If it does not help, your condition/disease may get worse.

You may have problems because of the drugs used in this study. These problems are called side effects. Some side effects are just bothersome. Others could harm you. There may be some side effects that we do not know about yet. The research might involve risks to you that are currently unforeseeable. Your study doctor may give you medicines to help lessen side effects. Many side effects go away soon after you stop taking the study drug. In some cases, side effects can be serious, long lasting, or may never go away. There may also be the risk of death.

#### HERE ARE THE KNOWN SIDE EFFECTS THAT COULD HAPPEN WITH AVADOMIDE:

Avadomide has been given to people with cancer. The side effects reported by people who have taken Avadomide are listed below according to how frequently they were reported.

Very common side effects (greater than a 10% chance this will happen)

- Fatigue (tiredness) and weakness
- Anemia (decreased counts of red blood cells, a type of blood cell that carries oxygen)
- Neutropenia (decreased counts of neutrophils, a type of white blood cell that helps to fight infection)
- Thrombocytopenia (decreased counts of platelets, a type of blood cell that helps the blood to clot)
- Decreased appetite
- Nausea
- Vomiting
- Diarrhea
- Constipation
- Rash
- Fever
- Infections, including respiratory tract infection and pneumonia (lung infection)

#### Common side effects (between 1% and 10% chance this will happen)

- Febrile neutropenia (decreased white blood cells that help to fight infection with fever), requiring hospitalization and additional treatment
- Severe infections including, urinary tract infection, and sepsis (blood stream infection) that could result in death.
- Swelling of disease-affected lymph nodes and tumor sites causing pain, fever, and/or abnormal laboratory values. This is called tumor flare and usually occurs in the first cycle of treatment. Most participants who developed swelling of disease-affected lymph nodes and tumor sites had mild to moderate symptoms and recovered; however, one event of tumor flare reaction was fatal.

#### Less Common but Serious:

Other events reported in participants with cancer which may or may not be related to the study drug included:

- Blood clots (in the legs, lungs, or brain)
- Inflammation of the lungs (making it difficult to breathe)
- Development or worsening of pain and changes in sensations in nerves (tingling, burning) and decreased sense of touch (neuropathy)
- Elevated liver laboratory test results (showing abnormal liver function)
- Elevated kidney laboratory test results (showing abnormal kidney function). This can also occur as part of tumor lysis syndrome which refers to metabolic abnormalities arising from rapid destruction of cancer cells. This is rare and was seen in diseases like acute leukemia and high-grade lymphomas.

Some people with cancer taking Avadomine have reported later developing other cancers (second new cancers that are diagnosed in participants following a prior diagnosis of a first cancer).

Severe allergic reaction (angioedema) was reported in one study participant, who developed face and airway swelling, requiring admission to the hospital and intensive treatment followed by full recovery.

Laboratory tests in a few participants showed increased troponin (a test showing possible effects on heart muscle); however, other heart tests (ECG and ECHO/MUGA) in these participants were normal and they had no symptoms. Troponin decreased when study drug was interrupted. Updated safety data suggests no causal relation of heart dysfunction with avadomide.

Avadomide has been given to animals to find out what side effects might be seen in people. The most frequent side effects seen in animals include:

- Decreased appetite
- Weight changes
- Dehydration
- Inflammation of the lining of the stomach and intestine
- Effects on eyes, including red eyes and swelling of the middle layer of the eye, which could result in impaired vision
- Increased blood creatinine and urea (blood tests showing bad effects on the kidneys)

To prevent possible effects on kidneys, good hydration is recommended (participants are advised to drink plenty of fluids). Effects to heart muscle have been detected in two animals that received the highest dose of the study drug, but not seen in any other study animals.

Pre-clinical studies show that Avadomide absorbs UV light. It is not yet known if Avadomide may make your skin or eyes more sensitive to sunlight. As a precaution, participants are advised to avoid prolonged exposure to natural or artificial sunlight (UVA/B) while taking Avadomide by wearing sun-protective clothes, applying effective sunblock to your skin, and by wearing sunglasses.

Please let your study doctor know all of your present and past diseases and allergies and any medication you may be taking including over-the-counter medications, vitamins, herbal, homeopathic or holistic medications or treatments, as well as foods and beverages containing grapefruit. This is important because a possible interaction with some medications, vitamins, and remedies may cause serious side effects, and/or may still be unknown.

Your study doctor will tell you if any additional measures are needed. All participants taking part in the study will be watched carefully for any side effects and you should report any changes in the way you feel or your health to your study doctor.

Other things may happen as well from taking the study drug that your study doctor can tell you about. The study doctor may give you something to make the sick feeling go away, or may stop giving you the study drug.

#### **Risks Associated with Pregnancy**

Avadomide has some similarities to thalidomide. Thalidomide is known to cause severe life-threatening human birth defects. Avadomide is therefore considered to have the potential to cause birth defects in humans. If Avadomide is taken during pregnancy, it may cause birth defects or death to an unborn baby. Women must not become pregnant while taking Avadomide.

In an animal study, the tubes in the testicles where sperm is made were affected in some male rats after 3 months of receiving Avadomide and it is not currently known if this effect is reversible. The female animals were not affected and these changes were also not found in males of the other animal species tested. For male participants, the short- and long-term effects of Avadomide on the ability to make sperm and get a woman pregnant are currently unknown and, normally, it can take approximately 2-3 months to make new sperm. The effects of Avadomide on human fertility are currently not known, therefore all family planning options and/or alternatives should be thoroughly discussed with your study doctor prior to participating in this study.

Prior to signing and dating this consent form, there is important information for you to know about the pregnancy risk precautions for this study, that a woman of childbearing potential must use two effective birth control methods (for example: birth control pills, condoms) at the same time or practice complete abstinence from sexual contact with a man beginning 28 days before starting study treatment, throughout the entire duration of study treatment including, during any dose interruptions, and for at least 28 days after the end of study treatment with Avadomide.

All male participants must practice complete abstinence from sexual contact or use a condom during sexual contact with a pregnant woman or a woman of childbearing potential throughout the entire duration of study treatment including during dose interruptions, and for at least 3 months after the end of study treatment with Avadomide, even if you have undergone a vasectomy.

Before you consent to participating in this study, you will be counseled on the full requirements of the pregnancy precautions within the Avadomide Information Sheet that you have received and must agree to follow.

Other than the participant, women who are able to become pregnant and men who are able to father a child should not touch or handle the Avadomide capsules or the powder they contain unless they are wearing gloves.

You must never share your study drugs with others. You must not breastfeed or donate blood while you are participating in this study, and for at least 28 days after the last dose of study drugs. You must not donate sperm or semen while you are participating in this study, and for at least 3 months after the last dose of study drugs.

#### HERE ARE THE KNOWN SIDE EFFECTS THAT COULD HAPPEN WITH NIVOLUMAB:

Nivolumab may cause one or more of the side effects listed below. This information is based on data from cancer participants in other clinical trials with nivolumab. In addition, there may be side effects that are not yet known that may occur. You should tell your study doctor or study nurse right away about any possible side-effects you experience.

<u>Very common side effects of nivolumab [greater than or equal to 1/10 or greater than or equal to 10%]</u> are:

- Diarrhea
- Fatigue
- Itching
- Rash

Common side effects of nivolumab [greater than or equal to 1/100 to less than 1/10 or greater than or equal to 1% to less than 10%] include:

- Abdominal pain
- Alkaline phosphatase increased: lab test result associated with liver or bone abnormalities
- ALT increased: lab test result associated with abnormal liver function
- Amylase increased: lab test result associated with pancreas inflammation
- AST increased: lab test result associated with abnormal liver function.
- Chills
- Constipation
- Cough
- Creatinine increased: lab test result associated with decreased kidney function
- Decreased appetite
- Dizziness
- Dry mouth
- Dry skin
- Fever
- Headache
- Increased blood sugar
- Inflammation of the colon
- Inflammation of the mouth
- Infusion related reaction
- Lipase increased: lab test result associated with pancreas inflammation
- Joint pain or stiffness
- Loss of color (pigment) from areas of skin
- Lung inflammation (pneumonitis see details below)
- Musculoskeletal pain
- Nausea
- Redness
- Shortness of breath
- Sodium levels in the blood are low
- Swelling, including face, arms, and legs

- Thyroid gland function decreased
- Thyroid gland function increased
- Thyroid stimulating hormone increased: lab test result associated with abnormal thyroid function
- Tingling, burning, numbness or weakness, possibly in arms, legs, hands and feet
- Vomiting

#### Uncommon side effects of nivolumab [greater than or equal to 0.1% to less than 1%] include:

- Adrenal gland function decreased
- Allergic reaction/hypersensitivity
- · Bilirubin (liver function blood test) increased
- Bronchitis (inflammation of the tubes that carry air to and from the lungs)
- Cranial nerve disorder (caused by damage or inflammation to certain nerves in the brain and may cause eye problems/disorders and/or palsy)
- Diabetes
- Dry eye
- Hair loss
- Heart rate increased
- Heart rhythm abnormal
- High blood pressure
- Hives
- Inflammation of the eye
- Inflammation of the kidney
- Inflammation of the pancreas
- Inflammation of the pituitary gland
- Inflammation of the stomach
- Inflammation of the thyroid gland
- Liver inflammation
- Low blood pressure
- Lung infiltrates, associated with infection or inflammation
- Pituitary gland function decreased
- Psoriasis (characterized by patches of abnormal, scaly skin)
- Renal failure
- Respiratory failure
- Upper respiratory tract infection
- Vertigo (feeling off balance which can lead to dizziness)
- Vision blurred

## Rare side effects of nivolumab [greater than or equal to 1/10,000 to less than 1/1,000 or greater than or equal to 0.01% to less than 0.1%] include:

- Anaphylactic reaction (severe allergic reaction)
- Damage to the protective covering of the nerves in the brain and spinal cord
- Diabetes complications resulting in excess blood acids and diabetic coma
- Erythema multiforme: skin inflammatory reaction
- Guillain-Barre syndrome, an autoimmune disorder associated with progressive muscle weakness or paralysis

- Inflammation of blood vessels
- Inflammation of the brain, potentially life-threatening or fatal
- Inflammation of the heart
- Muscle inflammation
- Myasthenic syndrome (neurologic syndrome characterized by muscle weakness) including myasthenia gravis, a nerve disease that may cause weakness of eye, face, breathing, and swallowing muscles.
- Polymyalgia rheumatica, an inflammatory disorder causing muscle pain and stiffness
- Rhabdomyolysis: muscle fiber released into the blood stream which could damage your kidneys
- Rosacea: acne-like skin condition resulting in redness of face
- Sarcoidosis, a disease involving abnormal collections of inflammatory cells (granulomas) in organs such as lungs, skin, and lymph nodes
- Stevens Johnson syndrome: a serious and potentially life-threatening inflammatory disorder of skin and mucous membranes, resulting in blistering and shedding of skin
- Toxic epidermal necrolysis: a serious and potentially fatal disease characterized by blistering and peeling of the top layer of skin resembling a severe burn
- Histiocytic necrotizing lymphadenitis or Kikuchi lymphadenitis: disorder of the lymph nodes which causes the lymph nodes to become enlarged, inflamed and painful, commonly affecting lymph nodes of the neck and possibly associated with fever or muscle and joint pains.
- Vogt Koyanagi Harada syndrome; a disease that affects the pigmented tissue; this
  may affect the eye leading to swelling, pain and/or blurred vision; the ear leading to
  hearing loss, ringing in the ears and/or the skin leading to loss of skin color.

**Lung Inflammation (pneumonitis)**: It is possible that nivolumab may cause inflammation of the tissues of the lung. This adverse effect has been reported in participants treated with nivolumab. While many participants with x-ray or CT abnormalities have not developed any symptoms, some participants have developed mild to severe symptoms and in rare cases, death has occurred as a result of their lung inflammation. Signs and symptoms of lung inflammation may include:

- Difficulty breathing
- Pain or discomfort while breathing
- Chest pain
- Cough
- Shortness of breath
- Increased rate of breathing
- Fever
- Low blood oxygen levels
- Fatigue

Your study doctor and study nurse will watch you closely for changes in your ability to breathe and for other signs or symptoms that might show you are developing this type of lung inflammation and will perform regular tests including physical exams, measurement of oxygen levels through non-invasive testing (for example, pulse oximeter), blood tests, chest x-rays and/or CT scans.

Complications, including fatal events, have occurred in participants who received allogenic hematopoietic stem cell transplantation (HSCT) after nivolumab.

### Please inform your study doctor or study nurse AT ONCE if you experience any of the following:

- Any new or increased shortness of breath;
- Any new or increased chest pain;
- · Any new or increased pain/difficulty while breathing;
- Any new or increased cough or any significant change in your type of cough; for example, any new or increased mucous or blood in your cough;
- Any change in the amount of oxygen you require;
- Any fever, fatigue, or other symptoms that occur at the same time as any changes to your breathing or other lung symptoms.

If you start to develop symptoms, your study doctor will ask you to return to the clinic for additional tests, which could include a physical exam, measurement of oxygen levels, blood tests, chest x-rays, and/or CT scans. You will be monitored very closely for changes in your overall lung symptoms; monitoring may require hospitalization. You may require specific treatment in order to control pneumonitis. You may also be seen by a special doctor called a pulmonologist, who has special training to be an expert in how lungs work.

Prolonged treatment with medicines that suppress inflammation, sometimes needed to manage the side effects of nivolumab, may lower your body's ability to fight off certain infections (such as opportunistic infections). These infections may require treatment with antibiotic or antifungal medications and may be fatal.

Ask the study doctor or study staff if you have questions about the signs or symptoms of any side-effects you read about in this consent form.

#### RISKS ASSOCIATED WITH STANDARD OF CARE OR ALTERNATIVE TREATMENT:

As with any medication there may be risks, known and unknown.

A more complete listing of side effects for other therapies may be available for you to review if you wish. Please talk with your study doctor about the risks of both these study drugs and any alternative methods of treatment that are available.

#### WHAT CAN HAPPEN IF I GET INJECTIONS OR INFUSIONS?

You will receive Nivolumab as an intravenous (IV) infusion, which means you will receive it directly into your vein. This may cause the following problems:

- Irritation of the vein; your skin near the vein could become warm, swell, hurt, or get red
- Damage to your vein
- Damage to the skin or tissue around the injection site
- A blood clot or an air bubble could form, which could block a blood vessel in another part of your body

Some of these problems could be very serious.

Over time, getting a lot of injections can cause a vein to become hard or scar, which can make it difficult to put a needle into the vein to give you a shot or take blood.

#### **COULD I HAVE AN ALLERGIC REACTION?**

Sometimes people have allergic reactions to drugs (which includes the iodine dyes often used with CT scans). If you have a very bad allergic reaction, you could die. Some things that happen during an allergic reaction are:

- Rash
- Having a hard time breathing
- Wheezing when you breathe
- Sudden drop in blood pressure
- Swelling around the mouth, throat, or eyes
- Fast pulse
- Sweating

You should get medical help and contact the study doctor or study staff if you have any of these or any other side effects during the study.

## IS THERE ANY RISK TO YOUR UNBORN CHILDREN IF YOU TAKE PART IN THIS STUDY? For Women:

If you are pregnant, you cannot participate in this study because there may be risks to you and your unborn baby that are currently unforeseeable, risks that we do not know about yet. Breastfeeding (nursing) mothers will not be included in this study since it is not known whether the drugs in this study will be passed on to the baby in mother's milk. If you are currently breastfeeding and wish to continue breastfeeding, your study doctor may recommend another treatment. The study doctor will perform a blood pregnancy test before the start of the study for women who are able to have a baby.

Tell the study doctor right away if:

- You are pregnant.
- You become pregnant.
- You are planning to become pregnant
- You are breastfeeding.

#### For Men and Women:

Whether you are a man or a woman, there may be risks to your unborn children. If you take part in this study, you must agree to use an effective method of birth control as discussed with your study doctor during the time that you are on this study and through 28 days after last dose of CC-122 or 5 months after the last dose of nivolumab; whichever is longer (for women) and through 3 months after the last dose of CC-122 or 7 months after last dose of nivolumab; whichever is longer (for men).

Examples of effective birth control methods include:

- Barrier methods (diaphragm, condoms, spermicidal)
- Hormonal methods (oral birth control pills, birth control patch, shots or injections)
- Implanted devices (devices such as the copper intrauterine device (IUD))

- Surgical sterilization (tubal ligation or vasectomy)
- Abstinence (no sexual intercourse)

Examples of non-effective birth control methods include:

- IUD progesterone T
- Progesterone-only "minipill"
- Female condom
- Natural family planning (rhythm method) or breastfeeding
- Fertility awareness
- Withdrawal
- Cervical shield

You should discuss the method of birth control which is best for you to use both during study treatment and for a period of time after study treatment.

Whether you are a woman or a man, you should tell your study doctor immediately if you become pregnant or if your partner becomes pregnant. Women who become pregnant during the study will have to leave the study. The study doctor or study staff may ask for information about the pregnancy and the birth of the baby. The study doctor or study staff may share this information with the sponsor and Advarra IRB (a group of people who review research studies to protect the rights and welfare of research participants).

Cancer treatment can affect fertility in both men and women, and it is important to understand the risks before starting therapy. Ask your study staff about fertility preservation before you begin study treatment. However, once you have started study treatment you should not donate or sell your eggs or sperm.

### COULD I HAVE ANY OTHER PROBLEMS WITH MY HEALTH IF I DO THIS RESEARCH STUDY?

It is possible that you could have problems and side effects of Nivolumab and Avadomide that nobody knows about yet, which include your melanoma condition getting worse or even death. If the study doctor learns any new information about these study drugs that might change your mind about continuing in the study, the study doctor or study staff will tell you about it. The study doctor will also tell you if new treatments become available for your condition.

#### What are the risks of giving blood for this study?

Needle sticks carry some risks such as fainting, bleeding, bruising, discomfort, dizziness, infection and/or pain at the puncture site.

#### What are the risks of having a biopsy done for this study?

Risks include pain, discomfort, soreness, redness, swelling, bleeding, bruising, and/or drainage at the biopsy site, abnormal wound healing, fever, infection, allergic reaction to the medication used to numb the skin over the biopsy site, and missed abnormal tissue requiring the need for another biopsy.

A biopsy procedure will involve removing a part of your tumor. A core needle biopsy is a percutaneous ("through the skin") procedure that involves removing small samples of tumor tissue using a hollow "core" needle. An "excisional" biopsy is a surgical procedure where an entire mass or abnormal area is removed. In all procedures, the area around the tumor will be

anesthetized with an injection to help ease the pain and a sample will be removed either by cutting it out or removing tissue through a hollow "core" needle. There may be some bruising, bleeding, and soreness. There is a risk of the biopsy site getting infected. You may also be given medicine to make you sleepy.

#### What are the risks of other invasive study procedures?

#### MRI

Magnetic resonance imaging (MRI) uses a magnet and radio waves to make diagnostic medical images of the body. There have been no ill effects reported from exposure to the magnetism or radio waves used in this test. However, it is possible that harmful effects could be recognized in the future. A known risk is that the magnet could attract certain kinds of metal. Therefore, we will carefully ask you about metal within your body, including medical implants, devices such as pacemakers and internal defibrillators, or certain dyes found in tattoos. We will also keep the examining room locked so that no one carrying metal objects can enter while you are in the scanner.

If there is any question about potentially hazardous metal within your body, you will not undergo the MRI. This may exclude you from participation in this research study. The MRI involves entering a large room in which a magnet is present. You will be placed on a narrow bed and then slid into a small tunnel approximately 6 feet in length and 25 inches in diameter. You will be asked to lie still for about one hour on this bed. You will hear a loud machine-like noise. You may be asked to have a harmless monitoring device applied during the MRI. During the MRI, you can have voice contact and physical contact with someone in attendance if you desire. Let the study doctor know if you have a fear of enclosed spaces.

#### CT Scan

Computed Tomography (CT) is a way to make x-ray images of the inside of the body. The CT scanner is a doughnut-shaped machine that uses x-rays to create computer pictures that show structures inside your body more clearly than regular x-ray pictures. During the procedure, a technologist will take you into the CT scan room where you will lie down on the patient table (usually on your back) inside of the CT machine. You should get comfortable because it is very important that you not move during certain parts of the test.

CT examinations differ depending on the part of your body being studied. For example, if your abdomen is being studied, a series of pictures will be taken from your lower chest to your lower pelvis. During the study, you will be asked to hold your breath so that the pictures will not be blurred. The machine will make some noise, and the table will move during the scan. Also, you may receive signals from the technologist or from the machine about your breathing. Before or during the study, you may be given an injection of a contrast liquid in your vein to allow the radiologist to obtain clearer images of your organs. If you have any discomfort during the test or after the injection, be sure to tell the technologist.

#### **FDG-PET scans**

There is a chance that you may experience discomfort, pain, or swelling at the site where the radiotracer (FDG) is injected. There is a slight risk of having an allergic reaction to the radiotracer. The amount of radiation from the radiotracer is small and will be gone from your body in a few hours.

You will be exposed to radiation from x-rays used for PET scans in this trial, and from the FDG, itself. The amount of radiation to your body from FDG is small and will be gone from your body in a few hours. There is always a risk of developing a new cancer from being exposed to any radiation, including the low levels of x-rays used for a PET scan. The risk is thought to be low compared to the benefit the test can provide about your disease. Radiation from each PET scan you receive is equivalent to about 3 years of normal background radiation.

Whether or not you are in this clinical trial, you will probably have CT scans and/or PET scans to help your regular doctor treat your melanoma condition. If you participate in this clinical trial, you may have more CT scans and/or PET scans than you would if you were not in a clinical trial.

#### **ECHO or MUGA**

If you have an ECHO, electrodes will be placed on your chest. You may feel some discomfort similar to pulling off an adhesive bandage when the technician removes the electrodes after the procedure. During a MUGA, a small amount of a radioactive chemical will be injected into your veins. The radiation exposure from this is considered small and is not likely to adversely affect you or your disease.

#### Confidentiality

There is a risk of loss of confidentiality of your information. You will read more about the protection of your information later in this form. Please ask the study doctor or study staff if you would like to know more about how your information will be protected while you are in this study.

#### WHAT IF I GET HURT OR SICK WHILE I AM IN THIS STUDY?

#### If you need emergency care:

 Call 911 or go to your nearest emergency room right away. Moffitt Cancer Center does not have an emergency room or the facilities to provide emergency care.

#### If you do NOT need emergency care:

Call or go to your regular doctor. It is important that you tell your regular doctor that you
are participating in a research study. If possible, take a copy of this consent form with
you when you go.

If you experience a side effect or a change in the way that you feel, call the study doctor at the telephone number listed on the first page of this form.

By signing this informed consent and research authorization form, you have not given up any legal rights to seek compensation for injuries from the sponsor.

#### MOFFITT CANCER CENTER INJURY STATEMENT

If you believe you have been injured as a result of your participation in this study or if you have questions about your rights as a person who is taking part in a research study, you may call the Moffitt Cancer Center Risk Manager at 813-745-7882. Moffitt Cancer Center and its investigators have made no provision for monetary compensation in the event of physical illness or injury resulting from this study. Likewise, Moffitt Cancer Center and its investigators have made no provision for payment of lost wages, disability, or discomfort in the event of physical illness or injury resulting from this study. Florida law (Statute 768.28) limits the liability of Moffitt Cancer Center. This statute provides that damages are available only to the extent that

negligent conduct of a Moffitt Cancer Center employee caused your injuries, and are limited by law. A copy of this statute is available upon request at 813-745-1869.

#### **WILL I GET PAID?**

You will not be paid for taking part in this research study. You have no rights to and will not receive payments of any kind for discoveries, patents or products that may be developed from this study.

#### WHILE YOU ARE IN THE STUDY, YOU MUST:

- Follow the instructions you are given.
- Come to the study center for all visits with the study doctor.
- Give correct and accurate information about your medical history and current medical condition.
- Tell the study doctor about any health problems you have during the study.
- Tell the study doctor about any new medicine or drug you take during the study.
- Not take any other drugs or remedies unless the study doctor has approved them beforehand. This includes prescription drugs and over the counter medicine (including vitamins and herbal remedies) that you buy without a prescription.
- Not participate in other medical research studies.
- Not get pregnant or cause your partner to become pregnant.
- Tell the study doctor or study staff if you want to stop being in the study at any time.

#### DO I HAVE TO REMAIN ON THIS STUDY ONCE I JOIN?

Your participation in this study is voluntary and you do not have to participate. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. Leaving the study will not affect your medical care. You can still get your medical care from our institution.

Tell the study doctor if you are thinking about stopping or deciding to stop. If you do decide to stop your participation in the study, your study doctor will tell you how to stop safely and will discuss with you what follow-up care or testing would be helpful to you. The study doctor may stop you from taking part in this study at any time if he/she believes it is in your best interest, if you do not follow the study rules, or if the study is stopped

## ARE THERE REASONS THE STUDY DOCTOR OR SPONSOR MIGHT TAKE ME OUT OF THE STUDY LATER?

Even if you want to stay in the study, there may be reasons the study doctor or study staff will need to take you out of it. Your study doctor has the right to take you out of the study at any time with or without your agreement. Your participation may be ended without your consent for different reasons, including the following:

- If the study doctor believes, for any reason, that it is in your best interest.
- If at any time while you are taking the study drug the study doctor discovers that your disease has worsened.
- If you develop side effects that the study doctor considers unacceptable.

- If you refuse to take the study drug or return for follow-up as recommended by your study doctor, or do not follow the study doctor's instructions.
- If you refuse to have tests that are needed to determine whether the study drug is safe and effective.
- If you require treatment with drugs that are not allowed on this study.
- If other causes prevent you from continuing in this study.
- If the Sponsor decides to end the study.

#### **HOW WILL MY INFORMATION BE KEPT CONFIDENTIAL?**

We understand that information about you and your health is personal, and we are committed to protecting the privacy of that information. Because of this commitment and because of federal law, we must obtain your written authorization before we use or disclose your information for this study.

By signing this form, you are permitting researchers at Moffitt Cancer Center to use personal health information for research purposes within its organized health care arrangements. You are also allowing the Moffitt Cancer Center to disclose your personal health information to outside organizations or individuals that participate in this study. We may publish what we find out from this study. If we do, we will not let anyone know your name. We will not publish anything that would directly let people know who you are.

#### WHO WILL DISCLOSE, RECEIVE, AND/OR USE YOUR INFORMATION?

Your records are confidential and they will be kept in a secure environment and protected to the full extent of the law.

To do this research, the following people and/or organization(s) will be allowed to disclose, use, and receive your information, but they may only use and disclose the information to the other parties on this list, to you or your personal representative, or as permitted by law:

- Every research site for this study, including the Moffitt Cancer Center, and each site's study team, research staff and medical staff.
- Any person who provides services or oversight responsibilities in connection with this study.
- Every member of the Moffitt Cancer Center workforce who provides services in connection with this study.
- The person who is responsible for the study nationwide or worldwide (study chairperson).
- Any laboratories, individuals, and organizations that use your health information in connection with this study.
- Any sponsor of the study, including the following sponsors: Moffitt Cancer Center, Celgene (funding the study), Bristol Myers Squibb (supplying study drug).
- Any federal, state, or local governmental agency that regulates the study (such as the U.S. Food and Drug Administration (FDA) and Florida Department of Health (FDH). The U.S. Department of Health & Human Services (DHHS), Office for Human Research Protections (OHRP).
- Other government agencies in this or other countries.

- The designated Protocol Review and Monitoring Committees, Institutional Review Boards such as Advarra IRB, Privacy Boards, Data and Safety Monitoring Board and their related staff that have oversight responsibilities for this study.
- The National Cancer Institute in evaluating the ongoing research of the Moffitt Cancer Center as a Comprehensive Cancer Center.

The organizations and people listed above may employ or pay various consultants and companies to help them understand, analyze and conduct this study. All of these people may not be known now, but if you would like to have more specific information about this at any time during the study, you may ask the study doctor and your questions will be answered.

Moffitt Cancer Center cannot guarantee the privacy of your information, or block further use or distribution, after the information has left the Moffitt Cancer Center. Others listed above may further disclose your information, and it may no longer be covered by federal privacy regulations. If all information that does or can identify you is removed from your records, the remaining information will no longer be subject to this authorization and may be used or shared for other purposes. You might have the right to see and copy your health records related to this research. You might not be able to see or copy some of your records until after all participants finish the study. If it is necessary for your care, your records will be provided to you or your regular doctor.

#### WHAT INFORMATION WILL BE USED OR DISCLOSED?

By signing below, you authorize the use and disclosure of your entire study record and any medical or other records held by Moffitt Cancer Center, including, but not limited to, HIV/AIDS, mental health, substance abuse or genetic information. The purpose for the uses and disclosures you are authorizing is to conduct the study explained to you during the informed consent and research authorization process and to ensure that the information relating to that study is available to all parties who may need it for research purposes.

Your authorization to use your health information will never expire unless and until you expressly revoke it in writing to the study doctor listed on the first page of this form.

Any data collected before your letter will continue to be used as necessary to preserve the integrity of the study, however no additional information will be collected after you withdraw your authorization.

You will receive a signed and dated copy of this form.

#### WHOM TO CONTACT ABOUT THIS STUDY

During the study, if you experience any medical problems, suffer a research-related injury, or have questions, concerns or complaints about the study, please contact the Investigator at the telephone number listed on the first page of this consent document. If you seek emergency care, or hospitalization is required, alert the treating physician that you are participating in this research study.

An institutional review board (IRB) is an independent committee established to help protect the rights of research participants. If you have any questions about your rights as a research participant, and/or concerns or complaints regarding this research study, contact:

By mail:

Study Participant Adviser Advarra IRB 6940 Columbia Gateway Drive, Suite 110 Columbia, MD 21046

• or call **toll free**: 877-992-4724

or by <u>email</u>: <u>adviser@advarra.com</u>

Please reference the following number when contacting the Study Participant Adviser: Pro00032422.

#### WHERE CAN I GET MORE INFORMATION?

You may call the National Cancer Institute's (NCI) Information Service at:

1-800-4-CANCER (1-800-422-6237).

Visit the NCI's Websites at:

- CancerTrials: comprehensive clinical trial information at: http://cancertrials.nci.nih.gov
- CancerNet: accurate cancer information including PDQ at: <a href="http://cancernet.nci.nih.gov">http://cancernet.nci.nih.gov</a>

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### **STATEMENT OF CONSENT**

| I have read this form and its contents were explained to me for the purposes listed above. All of my questions were ans receive a signed and dated copy of this form for my records | swered to my satisfaction. I will |
|---|---|
| Printed Name of Participant | |
| Signature of Participant | Date / Time |
| STATEMENT OF PERSON OBTAINING INFORMED CON AUTHORIZATION | ISENT / RESEARCH |
| I attest that the participant named above had enough time to opportunity to ask questions, and voluntarily agreed to be in | |
| Printed Name of Person Explaining Consent | |
| Signature of Person Explaining Consent | Date / Time |